CLINICAL TRIAL: NCT06591455
Title: A Single Center, Randomized Controlled, Pilot Study of Fenofibrate and Ursodeoxycholic Acid in the Treatment of Newly Diagnosed Primary Biliary Cholangitis
Brief Title: A Pilot Study of Fenofibrate and Ursodeoxycholic Acid in the Treatment of Newly Diagnosed Primary Biliary Cholangitis
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: Han Ying (Other)
Responsible Party: Sponsor-Investigator, Han Ying, Professor, Xijing Hospital of Digestive Diseases
Organization: Xijing Hospital of Digestive Diseases (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: KY20242282
Record Dates: First submitted 2024-09-07; First posted 2024-09-19 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-06

CONDITIONS: Primary Biliary Cholangitis (PBC)
MeSH Terms: conditions — Liver Cirrhosis, Biliary | interventions — Fenofibrate; Ursodeoxycholic Acid

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- fenofibrate (Experimental): fenofibrate 200mg/day
  Interventions: Drug: Fenofibrate
- UDCA (Active Comparator): UDCA 13-15mg/kg/day
  Interventions: Drug: UDCA (Ursodeoxycholic acid)

INTERVENTIONS:
Drug: Fenofibrate — Fenofibrate 200mg/day
  Arms: fenofibrate
Drug: UDCA (Ursodeoxycholic acid) — UDCA 13-15mg/kg/day
  Arms: UDCA

SUMMARY:
This study is a prospective, single center, randomized controlled, exploratory clinical trial aimed at evaluating the efficacy and safety of fenofibrate in newly diagnosed PBC subjects.

ELIGIBILITY:
Inclusion Criteria:

* Must have provided written informed consent
* Age 18-75 years;
* BMI 17-28 kg/m2
* Male or female with a diagnosis of PBC, by at least two of the following criteria:

  1. History of AP above ULN for at least six months;
  2. Positive AMA titers (>1/40 on immunofluorescence or M2 positive by enzyme linked immunosorbent assay (ELISA) or positive PBC-specific antinuclear antibodies;
  3. Documented liver biopsy result consistent with PBC.
* Not receiving UDCA treatment before enrollment, ALP>ULN

Exclusion Criteria:

* History or presence of other concomitant liver diseases.
* ALT or AST > 5×ULN, TBIL > 3×ULN.
* If female: known pregnancy, or has a positive urine pregnancy test (confirmed by a positive serum pregnancy test), or lactating.
* Allergic to fenofibrate or ursodeoxycholic acid.
* Taking hepatotoxic drugs (e.g., dapsone, erythromycin, fluconazole, ketoconazole, rifampicin) for more than 2 weeks within 6 months, and long-term hormonal users.
* Recurrent variceal bleeding, poorly controlled hepatic encephalopathy or refractory ascites.
* Patients with a history of severe cardiac, cerebrovascular, renal, respiratory disease or functional failure, and psychiatric disorders (including those due to alcohol and drug abuse).
* Creatinine >1.5×ULN and creatinine clearance <60 ml/min.
* Currently using statins (such as pravastatin, fluvastatin, and simvastatin), other fibrates (such as gemfibrozil and bezafibrate), and drugs structurally similar to fenofibrate (like ketoprofen).
* Planned to receive an organ transplant or an organ transplant recipient.
* Needing Liver transplantation within 1 year according to the Mayo Rick score.
* Any other condition(s) that would compromise the safety of the subject or compromise

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2024-09-14 (Actual); Primary Completion 2025-08-18 (Actual); Study Completion 2025-08-18 (Actual)

PRIMARY OUTCOMES:
Percentage of patients with biochemical response | 6 months
  The normalisation of Alkaline Phosphatase

SECONDARY OUTCOMES:
Percentage of patients having biochemical response | 1 and 3 months
  The normalisation of Alkaline Phosphatase
Assessment of the pruritus and fatigue | 1,3 and 6 months
  Change From Baseline in Fatigue and Pruritus as Assessed by Visual Analogue Scale (VAS) Total Score for Fatigue and Pruritus. (0-10, higher scires mean a worse outcome)

CONTACTS AND LOCATIONS:
Locations (1):
- Xijing hospital, Xi'an, Shaanxi, China